CLINICAL TRIAL: NCT01278784
Title: Local Tolerability of Chitosan-N-acetylcysteine Eye Drops in Healthy Young Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: OPHT-141010
Record Dates: First submitted 2010-12-20; First posted 2011-01-19 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye syndromes; Chitosan-N-Acetylcysteine
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy volunteer (Experimental)
  Interventions: Device: 0.05% Chitosan-N-Acetylcysteine eye drops; Device: 0.1% Chitosan-N-Acetylcysteine eye drops

INTERVENTIONS:
Device: 0.05% Chitosan-N-Acetylcysteine eye drops — Subjects will be randomized to receive one drop of the medical device in either the right or left eye
Device: 0.1% Chitosan-N-Acetylcysteine eye drops — Subjects will be randomized to receive one drop of the medical device in either the right or left eye

SUMMARY:
The "dry eye syndrome" DES is a highly prevalent ocular disease, in particular in the elderly population. One mainstay of therapy for patients suffering from DES is the use of topically administered lubricants. However, despite many efforts, no "ideal" formulation has yet been found.

Recently, Croma Pharma has introduced chitosan-N-acetylcysteine eye drops, designed for treatment of symptoms related to DES. Chemically, chitosan is a polycationic biopolymer with favourable biological properties such as high biocompatibility and low toxicity. Additionally, the new formulation comprises N-acetylcysteine, which has been used in ophthalmology because of its mucolytic properties for several years. Based on theoretical considerations, one can hypothesize that the new chitosan derivative may show an increased adhesion to mucins of the ocular surface and may therefore be particularly beneficial in reducing the symptoms associated with DES. We have recently shown in a phase I trial that single instillation of chitosan-N-acetylcysteine eye drops is well tolerated in young healthy subjects. However, due to the fact that intraocular pressure has been measured as one of the main safety variables, topical anesthesia was necessary. Thus, the data about local ocular discomfort after administration are limited. This trial seeks to investigate whether single instillation of chitosan-N-acetylcystein leads to ocular discomfort such as burning and stinging.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 45 years
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 6 dpt

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks preceding the study
* Abuse of alcoholic beverages
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Ametropia less than 6 dpt
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Difference between 0.05% and 0.1% Chitosan-N-Acetylcysteine eye drops | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria